CLINICAL TRIAL: NCT07379216
Title: Efficacy Evaluation Study of Vitamin C and Glutathione Liquid Sachet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-103-A
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Skin Condition; Anti-Oxidative Stress
Keywords: Vitamin C supplement; Glutathione supplement
MeSH Terms: conditions — Skin Diseases | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo sachet
- Vitamin C and Glutathione Liquid Sachet (Experimental)
  Interventions: Dietary Supplement: Vitamin C and Glutathione Liquid Sachet

INTERVENTIONS:
Dietary Supplement: Placebo sachet — consume 1 sachet of the test samples daily for 12 consecutive weeks
  Arms: Placebo sachet
Dietary Supplement: Vitamin C and Glutathione Liquid Sachet — consume 1 sachet of the test samples daily for 12 consecutive weeks
  Other Names: Lipo GLUTA-C
  Arms: Vitamin C and Glutathione Liquid Sachet

SUMMARY:
The objective of this study is to evaluate the effect of liquid vitamin C and glutathione supplements on human skin condition improvement and anti-oxidation.

DETAILED DESCRIPTION:
This study is a single-center, placebo-controlled, double-blinded, parallel human trial designed to evaluate the skin beauty and anti-oxidant effect of liquid vitamin C and glutathione supplements.

Healthy adult participants aged 18-65 years will be enrolled. Participants will be informed to consume test samples daily for 12 consecutive weeks. Skin measurement and self-assessment questionnaires will be conducted at baseline (before intake), after 4, 8 weeks, and 12 weeks of consumption. Fasting blood samples will be collected at baseline and after 12 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, aged 18-65 years old;
* Commitment not to use products having activity comparable with that of the product to be tested during the study period;
* Free of any dermatological or systemic disorder that would interfere with results.

Exclusion Criteria:

* Subject with obvious skin surface damage;
* Subject who had oral or topical medication which may affect skin condition within 1 month;
* Individuals with known allergies to cosmetics, medications, or foods (especially those allergic to legumes/soy);
* Pregnant or breastfeeding individuals;
* Received facial laser therapy, chemical peeling in the past 2 months.
* Individuals unwilling to allow publication or public disclosure of photographs taken as part of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-24 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The change of skin tone | Change from Baseline skin tone at 12 weeks
  Chroma Meter MM500 was utilized to measure face skin tone. Units: Individual Typology Angle (ITA°)
The change of visible spots | Change from Baseline visible spots at 12 weeks
  VISIA Complexion Analysis was utilized to measure visible spots on face. Units: the amount of detectable visible spots
The change of UV spots | Change from Baseline UV spots at 12 weeks
  VISIA Complexion Analysis was utilized to measure UV spots on face. Units: the amount of detectable UV spots

SECONDARY OUTCOMES:
The change of skin hydration | Change from Baseline skin hydration at 12 weeks
  Corneometer® CM825 (CK, Germany) was utilized to measure skin surface hydation. Units: arbitrary Corneometer® units 0-120.
The change of skin redness | Change from Baseline skin redness at 12 weeks
  Chroma Meter MM500 was utilized to measure face skin redness. Units: a* value
The change of skin melanin index | Change from Baseline skin melanin index at 12 weeks
  Mexameter® MX18 (CK, Germany) was utilized to measure face skin melanin level. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 12 weeks
  Skin elasticity (Softplus, Italy) was utilized to measure face skin elasticity. Units: arbitrary units
The change of brown spots | Change from Baseline brown spots at 12 weeks
  VISIA Complexion Analysis was utilized to measure brown spots on face. Units: the amount of detectable brown spots
The change of wrinkles around the eyes | Change from Baseline wrinkles around the eyes at 12 weeks
  VISIA Complexion Analysis was utilized to measure wrinkles around the eyes. Units: the amount of detectable wrinkles
The change of skin texture | Change from Baseline skin texture at 12 weeks
  VISIA Complexion Analysis was utilized to measure skin texture. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 12 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin collagen density. Units: arbitrary units
The change of total antioxidation capacity (TAC) | Change from Baseline TAC at 12 weeks
  A fasting blood sample will be collected for TAC testing.
The change of Superoxide Dismutase (SOD) | Change from Baseline SOD at 12 weeks
  A fasting blood sample will be collected for SOD testing.
The change of Glutathione S-transferase-Red Blood Cells (GST-RBC) | Change from Baseline GST-RBC at 12 weeks
  A fasting blood sample will be collected for GST-RBC testing.
The change of Malondialdehyde (MDA) | Change from Baseline MDA at 12 weeks
  A fasting blood sample will be collected for MDA testing.

OTHER OUTCOMES:
The change of self-assessment skin condition | Change from Baseline skin condition at 12 weeks
  Skin condition was evaluated using a 5-point Likert scale (0-4) to assess the severity of skin-related symptoms. The scale was defined as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
The change of self-assessment fatigue level | Change from Baseline fatigue level at 12 weeks
  Fatigue Symptom Inventory (FSI) was collected and evaluate fatigue level. Most items are rated on an 11-point Likert scale ranging from 0 to 10. The scores are generally averaged to create subscales for intensity and interference.
The change of self-assessment Low Immunity level | Change from Baseline Low Immunity level at 12 weeks
  Low Immunity level was evaluated using a 5-point Likert scale (0-4) to assess the severity of Low Immunity-related symptoms. The scale was defined as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
The change of blood liver function biomarkers (AST, ALT) | Change from Baseline liver function biomarkers at 12 weeks
  A fasting blood sample will be collected for liver function biomarkers testing.
The change of blood renal function biomarkers (creatinine, BUN) | Change from Baseline renal function biomarkers at 12 weeks
  A fasting blood sample will be collected for renal function biomarkers testing.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D., Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Pingtung City, Taiwan